CLINICAL TRIAL: NCT04101760
Title: Long-acting Versus Short-acting Granulocyte Colony Stimulating Factor for the Prevention of Febrile Neutropenia in Epithelial Ovarian Cancer Patients: A Multicenter Phase 3 Randomized Controlled Study
Brief Title: Granulocyte Colony Stimulating Factor for for the Prevention of Febrile Neutropenia in Epithelial Ovarian Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lei Li (Other)
Collaborators: Beijing Hospital (Other Government); China-Japan Friendship Hospital (Other); Navy General Hospital, Beijing (Other); Seventh Medical Center of PLA Army General Hospital (Other)
Responsible Party: Sponsor-Investigator, Lei Li, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EOC-CSF
Record Dates: First submitted 2019-09-21; First posted 2019-09-24 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Chemotherapy-induced Neutropenia; Febrile Neutropenia, Drug-Induced; Epithelial Ovarian Cancer; Colony Stimulating Factors Adverse Reaction; Granulocyte Colony Stimulating Factor; Cost-effectiveness Analysis; Quality of Life; Progression-free Survival; Overall Survival
MeSH Terms: conditions — Chemotherapy-Induced Febrile Neutropenia; Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Patients in study group accept prophylactic treatment of long-acting granulocyte colony stimulating factor
  Interventions: Drug: Long-acting granulocyte colony stimulating factor
- Control group (Active Comparator): Patients in control group accept regular or prophylactic treatment of short-acting granulocyte colony stimulating factor according to current guidelines
  Interventions: Drug: Short-acting granulocyte colony stimulating factor

INTERVENTIONS:
Drug: Long-acting granulocyte colony stimulating factor — Patients will accept long-acting granulocyte colony stimulating factor at 48 hour after the chemotherapy
  Arms: Study group
Drug: Short-acting granulocyte colony stimulating factor — Patients will accept short-acting granulocyte colony stimulating factor followed regular or prophylactic patterns
  Arms: Control group

SUMMARY:
This study aims to analyze the effects of long-acting versus short-acting granulocyte colony stimulating factor (G-CSF) on the prevention febrile neutropenia (FN) in epithelial ovarian cancer patients.

Patients receive platinum-based chemotherapy of 3 to 4 weeks. Patients are randomized into study group and control group. In study group, patients accept long-acting G-CSF 48 hours from the chemotherapy. While the control group accept regular or prophylactic treatment of short-acting G-CSF according to National Comprehensive Cancer Network guidelines.

The primary end is the incidence of FN in every course of chemotherapy.

The secondary ends include: the incidences of myelosuppression, doses of G-CSF and its expenses, visits to outpatient and emergency clinics, adverse events related to G-CSF, quality of life, and survival outcomes (progression-free survival and overall survival).

ELIGIBILITY:
Inclusion Criteria:

* With definitive pathological results of epithelial ovarian cancer
* With an Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2
* Aged 18 or older
* Receiving 3-4 weeks per cycle of platinum-based chemotherapy with or without debulking surgery
* Regularly followed up in the study centers
* Provided consent for participation.

Exclusion Criteria:

* Failure to meet all the inclusion criteria
* Non-compliance with the study protocols
* With a history of chemotherapy or pelvic radiotherapy for malignancies
* Presence of immunosuppressive diseases such as organ transplantation or acquired immune deficiency syndrome
* Treated with weekly chemotherapy regimens
* Presence of hematological disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of febrile neutropenia | One year
  Incidence of febrile neutropenia during each course of chemotherapy

SECONDARY OUTCOMES:
Incidence of myelosuppression | One year
  Incidence of febrile neutropenia during each course of chemotherapy
Doses of granulocyte colony stimulating factor | One year
  Doses of long-acting and short-acting granulocyte colony stimulating factor used during each course of chemotherapy
Numbers of visits to the hospital | One year
  Visits to the outpatient clinics and emergency room
Adverse events | One years
  Incidence of adverse events related to granulocyte colony stimulating factor according to Common Terminology Criteria for Adverse Events (CTCAE) v4.03
Progression-free survival | Two years
  Progression-free survival after the treatment of ovarian cancer during the study periods
Overall survival | Two years
  Overall survival after the treatment of ovarian cancer during the study periods

CONTACTS AND LOCATIONS:
Overall Officials: Lei Li, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Lei Li, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data will be shared as a supplement along with the published papers.
Supporting Information: Study Protocol